CLINICAL TRIAL: NCT03432286
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Galcanezumab in Patients 6 to 17 Years of Age With Episodic Migraine - the REBUILD-1 Study
Brief Title: A Study of Galcanezumab (LY2951742) in Participants 6 to 17 Years of Age With Episodic Migraine
Acronym: REBUILD-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16352; I5Q-MC-CGAS (Other: Eli Lilly and Company); 2017-004351-23 (EudraCT Number)
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Episodic Migraine
Keywords: pediatric; children; prevention; prophylaxis; headache; pediatric migraine
MeSH Terms: conditions — Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galcanezumab (Experimental): Galcanezumab administered by SQ injection.
  Participants may be eligible for optional open-label extension at the end of the double-blind period.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo administered by SQ injection.
  Participants may be eligible for optional open-label extension at the end of the double-blind period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SQ
  Other Names: LY2951742
  Arms: Galcanezumab
Drug: Placebo — Administered SQ
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaulate the efficacy and safety of galcanezumab in participants 6 to 17 years of age for the preventive treatment of episodic migraine. The primary objective is to demonstrate the superiority of galcanezumab versus placebo in the reduction of monthly migraine headache days across the 3-month double-blind treatment period.

DETAILED DESCRIPTION:
The study has two parts which enroll separately from each other such that participants may choose to participate in either but not both: the main study and a study addendum.

* The main study includes a 3-month, randomized, double-blind treatment period in which participants receive either galcanezumab or placebo, followed by a 9-month open-label extension in which all participants receive galcanezumab.
* The study addendum is a stand-alone study of galcanezumab pharmacokinetics and safety in a group of participants separate from those in the main study. The study addendum includes a 5-month evaluation period after a single injection of galcanezumab, followed by a 9-month open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine with or without aura as defined by the IHS ICHD-3 guidelines (1.1 or 1.2 according to ICHD-3 [2018]), with a history of migraine headaches of at least 6 months prior to screening.

Exclusion Criteria:

* Participants who are taking, or are expected to take, therapeutic antibodies during the course of the study (adalimumab, infliximab, trastuzumab, bevacizumab, etc.). Prior use of therapeutic antibodies is allowed if that use was more than 12 months prior to baseline.
* Known hypersensitivity to monoclonal antibodies or other therapeutic proteins, or to galcanezumab or its excipients.
* Current use or prior exposure to galcanezumab, another CGRP antibody, or CGRP receptor antibody, including those who have previously completed or withdrawn from this study or any other study investigating a CGRP antibody.
* History of IHS ICHD-3 diagnosis of new daily persistent headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine and migraine with brainstem aura (previously basilar-type migraine).
* History of significant head or neck injury within 6 months prior to screening; or traumatic head injury at any time that is associated with significant change in the quality or frequency of their headaches, including new onset of migraine following traumatic head injury.
* Participants with a known history of intracranial tumors or developmental malformations including Chiari malformations.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 533 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Number of Monthly Migraine Headache Days | Baseline, 3 Months
  Change from baseline in the number of monthly migraine headache days

SECONDARY OUTCOMES:
Percentage of Participants with Reduction from Baseline ≥50%, ≥75% and 100% in Monthly Migraine Headache Days | 3 Months
  Percentage of participants with reduction from baseline ≥50%, ≥75% and 100% in monthly migraine headache days
Change from Baseline in the Number of Monthly Migraine Headache Days with Nausea and/or Vomiting | Baseline, 3 Months
  Change from baseline in the number of monthly migraine headache days with nausea and/or vomiting
Change from Baseline in the Number of Monthly Migraine Headache Days with Photophobia and Phonophobia | Baseline, 3 Months
  Change from baseline in the number of monthly migraine headache days with photophobia and phonophobia
Change from Baseline in the Number of Monthly Migraine Headaches with Prodromal Symptoms | Baseline, 3 Months
  Change from baseline in the number of monthly migraine headaches with prodromal symptoms
Change from Baseline in the Number of Migraine Headache Days on which Acute Headache Medication is Taken | Baseline, 3 Months
  Change from baseline in the number of migraine headache days on which acute headache medication is taken
Patient Global Impression-Improvement (PGI-I) Rating | Month 1 to Month 3
  PGI-I rating
Change from Baseline in the Severity of Remaining Migraine Headaches per Month | Baseline, 3 Months
  Change from baseline in the severity of remaining migraine headaches per month
Change from Baseline in the Number of Monthly Headache Days | Baseline, 3 Months
  Change from baseline in the number of monthly headache days
Change from Baseline on the Pediatric Quality of Life Inventory (PedsQL) Total Score | Baseline, 3 Months
  Change from Baseline on the PedsQL total score
Change from Baseline on the Pediatric Migraine Disability Assessment Test (PedMIDAS) Total Score | Baseline, 3 Months
  Change from baseline on the PedMIDAS total score
Percentage of Participants with Suicidal Ideation and Behaviors Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Score | Baseline through 3 Months
  Percentage of Participants with Suicidal Ideation and Behaviors Assessed by the C-SSRS Score
Pharmacokinetics (PK): Serum Concentration of Galcanezumab | Baseline through 3 Months
  PK: Serum concentration of galcanezumab
Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP) | Baseline through 3 Months
  Plasma concentration of CGRP
Percentage of Participants Developing Anti-Drug Antibodies | Baseline through 3 Months
  Percentage of participants developing anti-drug antibodies
Percentage of Participants who Initiate Migraine Prevention Medication in the Post-Treatment Follow-Up Phase | 16 Months
  Percentage of participants who initiate migraine prevention medication in the post-treatment follow-up phase

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (73):
- United States (38):
  - Rehabilitation & Neurological Services, Huntsville, Alabama
  - 21st Century Neurology, a Division of Xenoscience, Inc., Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - Wr-McCr, Llc, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - University of Miami Don Suffer Clinical Research Building, Miami, Florida
  - Ezy Medical Research, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - USF Health, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Clinical Integrative Research Center of Atlanta, LLC, Atlanta, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Medical Research Partners, Ammon, Idaho
  - Elite Clinical Trials, Blackfoot, Idaho
  - Northwest Clinical Trials, Boise, Idaho
  - Inpatient Pharmacy, Hoffman Estates, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Minneapolis Clinic of Neurology - Burnsville Office, Burnsville, Minnesota
  - Children Mercy Pediatric Clinical Research Unit, Kansas City, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Cohen Children's Northwell Health Physician Partners - Pediatric Neurology, New Hyde Park, New York
  - Velocity Clinical Research at Raleigh Neurology, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Providence Health & Services, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Office 18, Pittsburgh, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Pain and Headache Centers of Texas, Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Children's Hospital, Seattle, Washington
- Denmark (2):
  - Sanos Clinic - Nordjylland, Aalborg
  - Herlev and Gentofte Hospital, Copenhagen
- Praxis Dr. Astrid Gendolla, Essen, Germany
- India (8):
  - Mangala Hospital & Mangala Kidney Foundation, Mangalore
  - Getwell Hospital and Research Institute, Nagpur
  - Central India Cardiology and Research Institute, Nagpur
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Medipoint Hospitals Pvt. Ltd., Pune
- Italy (3):
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Policlinico Umberto I, Roma
- Japan (8):
  - Konan Hospital, Kobe
  - Umenotsuji Clinic, Kochi
  - Tatsuoka Neurology Clinic, Kyoto
  - Yamaguchi Clinic, Nishinomiya
  - Tominaga Hospital, Osaka
  - Sendai Headache and Neurology Clinic, Sendai
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Tokyo Headache Clinic, Tokyo
- Mexico (5):
  - Centro de Investigacion Medica Aguascalientes (CIMA), Aguascalientes
  - Operadora Unidad de Investigación en Salud de Chihuahua S.A. de C.V., Chihuahua City
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
  - PanAmerican Clinical Research - Guadalajara, Guadalajara
  - Clinica De Enfermedades Cronicas y Procedimientos Especiales, Morelia
- Isala, locatie Zwolle, Zwolle, Netherlands
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC, Caguas
  - Ponce Medical School Foundation Inc., Ponce
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Galcanezumab (LY2951742) in Participants 6 to 17 Years of Age With Episodic Migraine — https://trials.lillytrialguide.com/en-US/trial/3ZYuzhkEA0eK8qoWk6AUq2